CLINICAL TRIAL: NCT03054246
Title: Chewing Side Preference is Associated With Hemispheric Laterality in Healthy Adults
Brief Title: Chewing Side Preference and Hemispheric Laterality in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Chewing side preference
Record Dates: First submitted 2017-02-09; First posted 2017-02-15 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Mastication

STUDY DESIGN:
Intervention Model Description: Healthy volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Other): Seventy-five healthy volunteers with no oral/dental problems with Angle I occlusion relationship and without any missing teeth will be included in the study. Evaluation of chewing side preference and laterality will be performed.
  Interventions: Other: Evaluation of chewing side preference

INTERVENTIONS:
Other: Evaluation of chewing side preference — The visual analog scale (VAS) is used. The individual will be asked to make 1 mark on a 10-cm line with " always left" and "always right" at either end and with " no preference" in the middle.

SUMMARY:
The study is aimed to investigate if chewing side preference (CSP) can be used as another indicator of hemispheric laterality in healthy adults. Healthy volunteers with no oral/dental problems with Angle I occlusion relationship and without any missing teeth will be included in the study. The CSP will be determined with the visual analog scale (VAS), which is the highly reliable method. Laterality test will be used to determine the preferred side for hands, feet, ears and eyes.

DETAILED DESCRIPTION:
Lateral preference is important to determine hemispheric laterality, which is usually diagnosed by hand and other sidedness, including footedness, eyedness and earedness. study is aimed to investigate if chewing side preference (CSP) can be used as another indicator of hemispheric laterality in healthy adults. Healthy volunteers with no oral/dental problems with Angle I occlusion relationship and without any missing teeth will be included in the study. The CSP will be determined with the visual analog scale (VAS), which is the highly reliable method. Laterality test will be used to determine the preferred side for hands, feet, ears and eyes.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers;

* Between the ages of 18-50 years
* Have no oral/dental problems with Angle I occlusion relationship and without any missing teeth
* Have no orofacial pain and/or no oral appliances will be included in the study.

Exclusion Criteria:

Participants;

* Under the age of 18 years and above the age of 50 years
* Have oral/dental problems with missing teeth
* Have orofacial pain
* Have oral appliances will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Chewing side | 1 month
  Evaluation of chewing side preference will be performed with VAS.

SECONDARY OUTCOMES:
Laterality | 1 month
  Evaluation of laterality will be performed with Laterality test

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serel Arslan S, Inal O, Demir N, Olmez MS, Karaduman AA. Chewing side preference is associated with hemispheric laterality in healthy adults. Somatosens Mot Res. 2017 Jun;34(2):92-95. doi: 10.1080/08990220.2017.1308923. Epub 2017 Apr 10. PMID 28393655